CLINICAL TRIAL: NCT05590130
Title: Comparison of Two Oxygenation Targets With Two Different Oximeters - Impact on Oxygen Flow Rates and Oxygenation
Acronym: Oxygap pong
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, François Lellouche, Principal investigator, Laval University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 22266
Record Dates: First submitted 2022-10-14; First posted 2022-10-21 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Oxygen Toxicity; Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Nonin oximeter with a 90% SpO2 target (Experimental): During this periods , oxygen will be administered in an manual titration with the FreeO2 device (fixed flow mode) to reach 90% of SpO2.
  Interventions: Device: Manual oxygen titration with Nonin oximeter (SpO2 target 90%)
- Philips oximeter with a 90% SpO2 target (Experimental): During this periods, oxygen will be administered in a manual titration with the FreeO2 device (fixed flow mode), to reach 90% of SpO2.
  Interventions: Device: Manual Oxygen titration with Philips oximeter (SpO2 target 90%)
- Nonin oximeter with a 94% SpO2 target (Experimental): During this periods , oxygen will be administered in a manual titration with the FreeO2 device (fixed flow mode) to reach 94% of SpO2.
  Interventions: Device: Manual oxygen titration with Nonin oximeter (SpO2 target 94%)
- Philips oximeter with a 94% SpO2 target (Experimental): During this periods, oxygen will be administered in a manual titration with the FreeO2 device (fixed flow mode), to reach 94% of SpO2.
  Interventions: Device: Manual Oxygen titration with Philips oximeter (SpO2 target 94%)

INTERVENTIONS:
Device: Manual Oxygen titration with Philips oximeter (SpO2 target 90%) — Oxygen titration with FreeO2 device (fixed flow mode) to reach the SpO2 target (set at 90%) with Philips oximeter
  Arms: Philips oximeter with a 90% SpO2 target
Device: Manual oxygen titration with Nonin oximeter (SpO2 target 90%) — Oxygen titration with FreeO2 device (fixed flow mode) to reach the SpO2 target (set at 90%) with Nonin oximeter
  Arms: Nonin oximeter with a 90% SpO2 target
Device: Manual Oxygen titration with Philips oximeter (SpO2 target 94%) — Oxygen titration with FreeO2 device (fixed flow mode) to reach the SpO2 target (set at 94%) with Philips oximeter
  Arms: Philips oximeter with a 94% SpO2 target
Device: Manual oxygen titration with Nonin oximeter (SpO2 target 94%) — Oxygen titration with FreeO2 device (fixed flow mode) to reach the SpO2 target (set at 94%) with Philips oximeter
  Arms: Nonin oximeter with a 94% SpO2 target

SUMMARY:
The investigators recently evaluated 4 different oximeters among the most commonly used with arterial catheter in place and compared SpO2 with SaO2 obtained on arterial gas. Correlations between SaO2 and SpO2 were poor for all oximeters, as previously known, and SpO2-SaO2 bias were different between oximeters. Some oximeters (Masimo, Nellcor) had lower biases but they detected less well hypoxemia. Some oximeters underestimated SaO2 (Nonin) but detected very well hypoxemia, and some overestimated SaO2 (Philips). The investigators concluded that oximeters provide different informations to clinicians, and oxygenation targets should take into account for these differences.

The assumption is that the SpO2 target AND oximeter used will both have an impact on oxygen flows and that these effects will add up. With a high SpO2 target, oxygen flows will be significantly greater and with the Nonin oximeter, the required flows will be greater than with the Philips oximeter.

NB: the results obtained were in a population with light skin pigmentation (96% of the patients were Fitzpatrick 1-2, reflecting the local hospitalized population).

DETAILED DESCRIPTION:
The oximeters to be evaluated will be the Nonin (Plymouth, MN), and the Philips (Eindhoven, Netherlands). The sensors used will be digital reusable sensors for all oximeters. Because of the impact of the fingers used for SpO2 measurement, each oximeter will be randomly assigned a different finger to each patient (digit 2 and 3 on the hand opposite to the arterial catheter).

Two SpO2 targets will be assessed: 90% and 94%. A total of four 10-minute periods will be performed in randomized order: Nonin 90, Nonin 94, Philips 90, and Philips 94.

At the end of each 10-minute period, arterial gas will be collected through the arterial catheter.

The adjustment of the oxygen flow rates will be performed manually. The average oxygen flow of the last 2 minutes of the period will be considered.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Patients admitted to postoperative cardiac surgery intensive care unit
* Presence of an arterial catheter Specific for the extubate patient
* Ongoing on conventional oxygen therapy at moderate flow (up to a maximum of 5L/min) with SpO2 between 88 and 100% with the usual oximeter and nasal cannula.
* SpO2 < 92% ambient air Specific for the intubate patient FiO2 <= 0.60 with SpO2 between 88 and 100% with usual oximeter SpO2 < 92% with FiO2 0.21

Exclusion Criteria:

* No SpO2 signal with oximeter in use
* False nails or nail polish
* Methemoglobinemia >0.015 on last available arterial gas
* Patient in isolation (multi-resistant bacteria, C-Difficile, SARS-CoV-2 ...) Specific for the extubate patient
* Expected to use another respiratory support within one hour of inclusion (NIV or nasal high flow oxygen) Planned extubation within one hour of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Oxygen flow (or FiO2) | Mean Oxygen flow in the two last minute of each study period (between minute 8 and 10)
  Oxygen flows (or FiO2) at the end of each study period (last minute average) to reach SpO2 target to reach SpO2 target with specific oximeter

SECONDARY OUTCOMES:
Difference between SpO2 and SaO2 | assessed up to 10 minutes - at the same of the arterial blood gases punction
  Difference (%) between SpO2 from each oximeter and SaO2 (% of SaO2 overestimation and underestimation for each oximeter)

OTHER OUTCOMES:
Mean difference on oxymeter | assessed up to 10 minutes - at the same of the arterial blood gases punction
  Mean (±SD) of the gaps between the different oximeters tested
Occult hypoxemia | assessed up to 10 minutes - at the same of the arterial blood gases punction
  Percentage of occult hypoxemia (SaO2<90% and SpO2>=90%)
Occult hyperoxemia | assessed up to 10 minutes - at the same of the arterial blood gases punction
  Perrcentage of occult hyperoxemia (SaO2>96% and SpO2<=96%)
Partial oxygen weaning | Mean oxygen flow in the two last minute of each study period (between minute 8 and 10)
  Rate of partial oxygen weaning (Oxygen flow <=0.5 L/min)
Complete oxygen weaning | Mean oxygen flow in the two last minute of each study period (between minute 8 and 10)
  Rate of complete oxygen weaning (Oxygen flow =0 L/min or FiO2 0.21)
Respiratory support escalation | Mean oxygen flow in the two last minute of each study period (between minute 8 and 10)
  Indication of initiation of respiratory support escalation (Oxygen flow >6 L/min or FiO2 > 0.60)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No